CLINICAL TRIAL: NCT02820779
Title: New Covered Stent (Willis) for the Endovascular Reconstruction of Intracranial Vessel Wall Defects Registry
Acronym: COVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: First Affiliated Hospital of Harbin Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Qilu Hospital of Shandong University (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Nanfang Hospital, Southern Medical University (Other); Tang-Du Hospital (Other); West China Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Shaanxi Provincial People's Hospital (Other); Shandong Provincial Hospital (Other Government); First Affiliated Hospital of Xinjiang Medical University (Other)
Responsible Party: Principal Investigator, Hongqi Zhang, MD, Cerebrovascular Expert Committee of Chinese Medical Doctor Association, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVER 001
Record Dates: First submitted 2016-06-23; First posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Aneurysm, Intracranial; Carotid-Cavernous Sinus Fistula
Keywords: Willis; Intracranial aneurysms
MeSH Terms: conditions — Intracranial Aneurysm; Carotid-Cavernous Sinus Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WILLIS (Experimental): Patients undergo WILLIS intracranial covered stent interventional treatment
  Interventions: Device: WILLIS

INTERVENTIONS:
Device: WILLIS — WILLIS® intracranial stent graft system is composed of the stent, delivery system, cobalt-based alloy stent and PTFE graft. It can effectively shunt the blood flow and keep it off of the aneurysm wall.
  Other Names: WILLIS® intracranial stent graft system

SUMMARY:
The purpose of this study is to evaluate the effectiveness, long-term safety and explore the safety and efficacy factors WILLIS™ intracranial stent graft system in clinical applications.

DETAILED DESCRIPTION:
Intracranial aneurysm is a cerebrovascular disorder in which weakness in the wall of a cerebral artery or vein causes a localized dilation or ballooning of the blood vessel.WILLIS® intracranial stent graft system is indicated for the treatment of intracranial aneurysms.

This study is a multi-center, prospective registration study.

Recruiting 100 specific patients to undergo a treatment with the WILLIS intracranial stent graft system, while giving the anti-platelet aggregation drugs and other medical therapy.

Patients enrolled will undergo a one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18;
* Arterial wall defects conformed by imaging examination due to internal carotid artery, vertebral artery aneurysms or various causes;
* Target lesion vessel reference diameter 3.5-4.5mm;
* Investigators believe that the patient is suitable for the interventional therapy of WILLIS intracranial covered stent;
* Participate in the study voluntarily, accept follow up study and signed Informed Consent Form.

Exclusion Criteria:

* Existence of branch artery (eg anterior choroidal artery, posterior communicating artery, posterior inferior cerebellar artery, etc.) of target lesion which may cause severe neurological dysfunction after occlusion;
* No suitable vessel entrance, or diseased artery extremely tortuous;
* Coagulation disorders or serious heart, liver, kidney dysfunction or systemic infection, which not suitable for interventional treatment;
* Life expectancy <1 year;
* Contraindications to heparin, aspirin, clopidogrel, anesthesia, X-ray or contrast agents;
* Mental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
1-year treatment success rate | 12 months
  Treatment success is defined as target lesion such as aneurysms, cavernous fistula shows no shadow and target vessel stenosis of no more than 50%.

SECONDARY OUTCOMES:
Technically success rate of surgery | immediately after surgery
  Technically success is defined as stent reach the target lesion and successfully released.
Target lesion treatment success rate | Immediately after surgery
X-ray exposure time | 24 hours
Operative time | through surgery completion
Surgery-related complications or death | 12 months
Various causes of death | the perioperative period to 12 months
Recurrence of target lesion | 12 months
Target lesion was treated by interventional or surgical therapy once again | 12 months
Postoperative ipsilateral symptomatic stroke | 30 days; 6 months; 12 months
  Ipsilateral symptomatic stroke is defined as the target lesion is conformed occurs ipsilateral stroke and the increase of NIHSS score point ≥4.
Occurs intracranial hemorrhagic stroke that caused by aneurysm rupture | 12 months
Occurs intracranial ischemic stroke that caused by thrombus | 12 months
All adverse events | 12 months
Device-related serious adverse events | 12 months
Target lesion appears stenosis 12 months after surgery | 12 months
  Stenosis is defined as target stenosis ≥50%
Modified Rankin Scale | 30 days; 6 months; 12 months
NIHSS | 30 days; 6 months; 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongqi Zhang, MD, Principal Investigator — hqzh@vip.163.com
Locations (11):
- China (11):
  - Nanfang hospital, Southern Medical university, Guangzhou, Guangdong
  - The 2nd Affiliated Hospital of Harbin Medical university, Harbin, Heilongjiang
  - The First Affiliated Hospital of Harbin Medical university, Harbin, Heilongjiang
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Qilu Hospital Of Shang Dong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - ShanXi Provincial People's Hospital, Taiyuan, Shanxi
  - Tangdu Hospital Fourth Military Medical University, Xi’an, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital Of Xinjiang Medical University, Ürümqi, Xinjiang
  - Tongji Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided